CLINICAL TRIAL: NCT03969264
Title: Tree Nut Consumption to Reduce Abdominal Adiposity and Risk for Metabolic Syndrome in Millennials
Brief Title: Tree Nut Consumption to Reduce Abdominal Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: International Tree Nut Council Research and Education Foundation (Unknown)
Responsible Party: Principal Investigator, Heidi J. Silver, Research Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VUMC71426
Record Dates: First submitted 2019-05-23; First posted 2019-05-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Millenials; Risk for Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized parallel two-arm study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and research assistant are blinded to study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carb Snacks (Active Comparator): Will follow study diet based on the Dietary Guidelines and consume study carbohydrate snacks between meals.
  Interventions: Other: High Carbohydrate or Tree Nut Food Snacks
- Tree Nut Snacks (Experimental): Will follow study diet based on the Dietary Guidelines and consume study tree nut snacks between meals.
  Interventions: Other: High Carbohydrate or Tree Nut Food Snacks

INTERVENTIONS:
Other: High Carbohydrate or Tree Nut Food Snacks — Snack consumption

SUMMARY:
A major contributing factor to the rising waist circumference of U.S. young adults is the increase in snacking behavior. Both the frequency of snacking during the day and the percentage of adults who engage in snacking has risen; national data indicates snacking comprises 15-25% of the total daily caloric intake of young and middle-aged adults. The overarching hypothesis, based on significant preliminary data, is that the quantity and metabolic function of abdominal fat is a key intermediary factor by which greater tree nut consumption reduces ectopic lipid storage (including the accumulation of intra-abdominal [visceral] fat), improves fatty acid and lipoprotein metabolism, reduces systemic inflammation and insulin resistance, and thus, reduces risk for MetS in millennial-generation age individuals.

DETAILED DESCRIPTION:
A major contributing factor to the rising waist circumference of U.S. young adults is the increase in snacking behavior. Both the frequency of snacking during the day and the percentage of adults who engage in snacking has risen; national data indicates snacking comprises 15-25% of the total daily caloric intake of young and middle-aged adults. Unfortunately, current typical snack items are energy rich, providing high intake of carbohydrates and sugars, as opposed to nuts that are nutrient rich. In prior work with middle-aged adults, the investigators found that consuming tree nuts daily as between-meal snacks for a period of 16 weeks significantly reduced intra-abdominal (visceral) fat and waist circumference, which was associated with altered plasma fatty acid profiles and higher fatty acid oxidation rates. Based on prior findings, the investigators propose to determine whether consuming mixed tree nuts as replacement for typical high carbohydrate snacks reduces abdominal obesity and waist circumference in millennials at risk for MetS. The overarching hypothesis, based on significant preliminary data, is that the quantity and metabolic function of abdominal fat is a key intermediary factor by which greater tree nut consumption reduces ectopic lipid storage (including the accumulation of intra-abdominal [visceral] fat), improves fatty acid and lipoprotein metabolism, reduces systemic inflammation and insulin resistance, and thus, reduces risk for MetS in millennial-generation age individuals. The hypothesis will be tested by determining: 1) the effect of consuming mixed tree nuts as daily snacks for 16 weeks on waist circumference and the quantity of abdominal fat (subcutaneous and visceral fat); 2) the effect of consuming mixed tree nuts as daily snacks for 16 weeks on circulating fatty acid profiles, glucose tolerance and insulin resistance, circulating lipids and lipoproteins, and circulating markers of inflammation; and 3) the effect of consuming mixed tree nuts as daily snacks for 16 weeks on abdominal tissue expression of genes that regulate inflammation, insulin resistance, and cardiometabolic mediators of MetS risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-36 years
* BMI 18.5 to 34.9
* At least one risk factor for metabolic syndrome based on waist circumference, HDL level or triglyceride level

Exclusion Criteria:

* Tree nut allergy
* Diagnosed chronic disease
* Medication for dyslipidemia or hypertension
* Smoke
* Weight loss medication
* Narcotic medication or illicit drug use
* Pregnancy or lactation or postmenopausal

Ages: 22 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 18 weeks
  Change in waist circumference (in centimeters)
Visceral Fat | 18 weeks
  Change in quantity of intra-abdominal fat by CT scan

SECONDARY OUTCOMES:
Gene Expression in Adipose Tissue | 18 weeks
  Change in expression of genes involved in regulation of inflammation and insulin resistance
Inflammation | 18 weeks
  Change in CRP level (mg/dl)
Dietary Macronutrient Intake | 18 weeks
  Change in macronutrient composition of the diet
Glucose | 18 weeks
  Change in fasting blood glucose (mg/dl)
Insulin | 18 weeks
  Change in serum insulin (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Silver, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD with other researchers.

REFERENCES:
- [Derived] Widmer A, Lillegard K, Wood K, Robles M, Fan R, Ye F, Koethe JR, Silver HJ. Consumption of tree nuts as snacks stimulates changes in plasma fatty acid profiles and adipose tissue gene expression in young adults at risk for metabolic syndrome. Clin Nutr. 2025 May;48:25-34. doi: 10.1016/j.clnu.2025.03.002. Epub 2025 Mar 8. PMID 40117963